CLINICAL TRIAL: NCT04268888
Title: A Two-arm Multi-stage (TAMS) Seamless Phase II/III Randomised Trial of Nivolumab in Combination With TACE/TAE for Patients With Intermediate Stage HCC
Brief Title: Nivolumab in Combination With TACE/TAE for Patients With Intermediate Stage HCC
Acronym: TACE-3
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Analysis meant the study should close to recruitment
Sponsor: The Clatterbridge Cancer Centre NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-9Y9
Record Dates: First submitted 2019-06-05; First posted 2020-02-13 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Intermediate Stage
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Patients shall be randomised on a 1:1 basis throughout the study and allocated using pre-generated lists produced by the study statistician. List shall be produced using permuted blocks algorithm with random block sizes of 2 and 4. Stratification factors used in the study are randomising centre, baseline HAP score (A vs. B vs. C) and vascular invasion (No vs. Yes).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TACE/TAE Alone (Active Comparator): Transarterial Chemoembolisation (TACE) and/or Transarterial Embolisation (TAE) Alone.
  Interventions: Procedure: TACE/TAE
- TACE/TAE and Nivolumab (Experimental): As above for TACE/TAE. Nivolumab adminstered as a flat dose of 480mg IV.
  Interventions: Drug: Nivolumab and TACE/TAE; Procedure: TACE/TAE

INTERVENTIONS:
Drug: Nivolumab and TACE/TAE — Immunotherapy and TACE/TAE
  Arms: TACE/TAE and Nivolumab
Procedure: TACE/TAE — TACE/TAE (as per local practice)

SUMMARY:
This study evaluates the addition of nivolumab to TACE/TAE in the treatment of patients with intermediate stage hepatocellular carcinoma. All patients will receive TACE/TAE and half will receive nivolumab.

DETAILED DESCRIPTION:
A significant proportion of HCC patients present with, or progress to, intermediate stage disease and these patients are typically treated with transarterial chemo-embolisation (TACE) or transarterial embolisation (TAE).

However, since TACE/TAE is generally a palliative therapy, it provides a potential backbone for the addition of effective systemic therapies with the aim of improving survival outcomes. Since TACE may liberate an abundance of tumour antigens and 'danger' signals, it may lend itself to combination with immunotherapeutic strategies.

Nivolumab is a human monoclonal antibody. Nivolumab targets the programmed death-1 PD-1) cluster of differentiation 279 (CD279) cell surface membrane receptor. PD-1 is a negative regulatory molecule expressed by activated T and B lymphocytes.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of HCC and at least one uni-dimensional lesion measurable according to RECIST 1.1 criteria by CT-scan or MRI.
2. Not a candidate for surgical resection or liver transplantation
3. Aged ≥16 years and estimated life expectancy >3 months
4. ECOG performance status 0-1
5. Adequate haematological function:

   * Hb ≥9g/L
   * Absolute neutrophil count ≥1.0x109/L
   * Platelet count ≥60x109/L
6. Bilirubin ≤50 μmol/L, AST,ALT and ALP ≤5 x ULN
7. Adequate renal function; Creatinine ≤ 1.5ULN (Using Cockcroft-Gault Formula)
8. INR ≤1.6
9. Child-Pugh A (score ≤6) (Appendix D)
10. HAP score A, B or C (Appendix E)
11. No contra-indications to T-cell checkpoint inhibitor therapy (use of immunosuppressive drugs including steroids at dose equivalent to prednisolone >10mg/day unless used as replacement therapy; organ transplantation; subjects with an active, known or suspected autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, lichen planus or other conditions not expected to recur in the absence of an external trigger are permitted to enrol).
12. Women of child-bearing potential should have a negative pregnancy test prior to study entry. Both men and women must be using an adequate contraception method, which must be continued for 5 months after completion of treatment for women and 7 months for men
13. Written informed consent

Exclusion Criteria:

1. Extrahepatic metastasis
2. Prior embolisation, systemic or radiation therapy for HCC
3. Any contraindications for hepatic embolisation procedures including portosystemic shunt, hepatofugal blood flow, known severe atheromatosis
4. Investigational therapy or major surgery within 4 weeks of trial entry
5. History of variceal bleeding within the past 4 weeks
6. Child-Pugh cirrhosis B or C (score ≥7)
7. HAP score D
8. Hepatic encephalopathy
9. Ascites refractory to diuretic therapy
10. Documented occlusion of the hepatic artery or main portal vein5
11. Hypersensitivity to intravenous contrast agents
12. Active clinically serious infection > Grade 2 NCI-CTC
13. Pregnant or lactating women
14. Known history of HIV infection
15. HBV chronic infection with HBV DNA > 500IU/mL or without antiviral therapy; HBV patients with cirrhosis should be treated.

17. History of second malignancy except those treated with curative intent more than three years previously without relapse and non-melanotic skin cancer or cervical carcinoma in situ 18. Evidence of severe or uncontrolled systemic disease, or laboratory finding that in the view of the Investigator makes it undesirable for the patient to participate in the trial 19. Psychiatric or other disorder likely to impact on informed consent 20. Patient is unable and/or unwilling to comply with treatment and study instructions 20. Interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected treatment-related pulmonary toxicity

21. Evidence of uncontrolled, active infection, requiring parenteral anti-bacterial, anti-viral or antifungal therapy within 7 days prior to administration of study medication

22. Positive test for latent TB or evidence of active TB

23. Hypersensitivity to any of the active substances or excipients

24. Patients who have received a live vaccine within 30 days prior to the first dose of trial treatment

25. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of the first dose of study drug administration

26. Any uncontrolled inflammatory GI disease including Crohn's Disease and ulcerative colitis

27. Participants with an active, known or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enrol

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 522 (Estimated)
Dates: Start 2019-05-08 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival - phase III primary outcome | The time until death. Patients discontinuing the study, lost to follow-up or still alive at the end of the study will be censored at the last know date alive, this can be assessed up until 2 years after the last patient.
  Measured in days
Time to TACE Progression (TTTP) - phase II primary outcome | The time to confirmatory scan 4 weeks after progression this can be assessed up until 2 years after the last patient is randomised
  Measured in days

SECONDARY OUTCOMES:
Time to Progression | Time to date of progression confirmed by RECIST1.1 assessed up until 2 years after the last patient is randomised
  Measured in days
Radiological response rate | Through study completion
  RECIST 1.1
Safety and Toxicity: the number and percentage of patients reporting a Serious Adverse Event (SAE) and Grade 3 or higher Adverse Event (AE) | Through study completion
  the number and percentage of patients reporting a Serious Adverse Event (SAE) and Grade 3 or higher Adverse Event (AE), measured and categorised based on CTCAE (version 4).
Progression Free Survival | Time to progression or death. Assessed up until 2 years.
  Measured in days
QOL: EORTC QLQ-C30 | baseline, pre - TACE (first treatment) and 12 weekly thereafter until end of treatment. Assessed up until 2 years after the last patient is randomised
  QoL will be scored according to the EORTC QLQ-C30 manual and guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Palmer, PhD, MD, Study Director — Clatterbridge Cancer Centre
Locations (2):
- Unicancer, Paris, France
- University of Liverpool, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kloeckner R, Galle PR, Bruix J. Local and Regional Therapies for Hepatocellular Carcinoma. Hepatology. 2021 Jan;73 Suppl 1:137-149. doi: 10.1002/hep.31424. Epub 2020 Nov 6. No abstract available. PMID 32557715